CLINICAL TRIAL: NCT04411173
Title: Effect of Daily Doses of Rice or Whey Protein on Resistance Training Adaptations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lindenwood University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: IRB-19-L0043
Record Dates: First submitted 2020-05-22; First posted 2020-06-02 (Actual); Last update posted 2020-06-02 (Actual); Status verified 2020-05

CONDITIONS: Hypertrophy
MeSH Terms: conditions — Hypertrophy | interventions — Whey Proteins

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: The supplements were delivered in identical containers with rather an "A" or "B" marked on the outside of the bag. Once data collection, data entry, and statistical analysis was completely finished, the study code was broken.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rice Protein (Active Comparator): Rice Protein - 24 grams, chocolate, powder
  Interventions: Dietary Supplement: Whey Protein
- Whey Protein (Active Comparator): Whey Protein - 24 grams, chocolate, powder
  Interventions: Dietary Supplement: Whey Protein

INTERVENTIONS:
Dietary Supplement: Whey Protein — Each condition (both rice and whey protein) match in color, flavor, and serving size.
  Other Names: Rice Protein

SUMMARY:
The purpose of this study is to compare the ability of isocaloric and isonitrogenous (2 x 15-gram) doses of rice protein or whey protein to stimulate resistance training adaptations in young, healthy, resistance-trained men.

DETAILED DESCRIPTION:
The study will be conducted using a randomized, double-blind approach with individuals being provided two doses of either 15 grams of rice or 15 grams of whey protein over an 8-week supplementation period while completing a heavy resistance training. One dose will be ingested within one hour of completing each workout and the other dose will be ingested within an hour of going to bed. On non-workout days, one dose of 30 grams will be ingested within 60 minutes of going to bed. The resistance training protocol will follow a linear periodization, split-body resistance training design consisting of two upper body and two lower body workouts each week resulting in each muscle group being trained twice each week. To minimize the influence of training experience and any learning effect, individuals with at least 12 months of resistance training history will be recruited. Participants will also be required to complete a two-week lead-in period (8 total workouts) before beginning the supplementation regimen to become accustomed to the training program and to account for any early neurological adaptations. Participants will then continue to follow the resistance training program for an additional 8 weeks. To assess the efficacy of the two different forms of protein supplementation on resistance training adaptations, changes in fat-free, lean, and fat mass will be determined using DEXA. Maximal strength and endurance of both upper and lower-body muscle groups will be determined while anaerobic capacity markers will be measured with the completion of a Wingate anaerobic capacity test. Participants will also be provided nutritional recommendations in order to ensure adequate energy and macronutrient consumption to facilitate positive training adaptations and eliminate any potential influence of differing dietary intakes.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18-50 years, although it is anticipated that the majority of participants will be between 18 and 35 years of age.
* Participants will be healthy and free of disease as determined by evaluation of a medical history
* All participants will be required to abstain from taking any additional forms of nutritional supplementation (preworkouts, creatine, beta-alanine, etc.) for four weeks prior to beginning this study and for the entire duration of the study.

Exclusion Criteria:

* Those individuals with less than 12 months of structured resistance training experience will be excluded from the study.
* Individuals whose maximal relative upper body strength is below 1.0 will be excluded.
* Individuals whose maximal relative lower body strength is below 1.50 will be excluded.
* As indicated on a medical history form they complete, any individual who is currently being treated for or diagnosed with a cardiac, respiratory, circulatory, musculoskeletal, metabolic, obesity (defined as body mass index > 30 kg/m2 and body fat greater than 30%), immune, autoimmune, psychiatric, hematological, neurological or endocrinological disorder or disease will be excluded.
* Those individuals who present with any previous injury or illness that would prevent them from appropriately completing all exercise lifts will be excluded from the study.
* Participants who are not able to fit onto the DEXA table will not be able to participate in the research due to size restrictions of the equipment. This typically includes individuals exceeding 300 pounds or those greater than 6 feet 6 inches.
* Those individuals less than 18 and greater than 50 years of age will be excluded. Participants younger than 18 are excluded due to necessity of parental consent. Participants greater than 50 years old lie outside of the target demographic for the current study.
* Participants who are determined to not be weight stable defined as week 0 and week 2 body mass levels deviating by 2% or more.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2018-09-12 (Actual); Primary Completion 2020-02-12 (Actual); Study Completion 2020-02-12 (Actual)

PRIMARY OUTCOMES:
Changes in upper- and lower-body strength via Dual-Energy X-ray Absorptiometry | Eight weeks
  Examining how much strength each participant gains (or loses) from Day 1 to Final day
Changes in fat-free mass via Dual-Energy X-ray Absorptiometry | Eight weeks
  Examining the differences in fat-free mass from Day 1 to Final day

SECONDARY OUTCOMES:
Changes in muscular endurance by counting repetitions for each exercise test | Eight weeks
  Examining the differences in muscular endurance from Day 1 to Final day
Changes in resistance training volume by tracking how many pounds were lifted during each exercise | Eight weeks
  Examining the differences in resistance training volume from Day 1 to Final day

CONTACTS AND LOCATIONS:
Overall Officials: Chad Kerksice, PhD, Study Director — Laboratory Director
Locations (1):
- Lindenwood University, Saint Charles, Missouri, United States

IPD SHARING:
Plan to Share IPD: No
All approved unidentified study data inside the laboratory will be saved within a research repository bank for future research questions. Otherwise, participant data will be destroyed after three years of study completion to maintain IRB compliance.

REFERENCES:
- [Derived] Moon JM, Ratliff KM, Blumkaitis JC, Harty PS, Zabriskie HA, Stecker RA, Currier BS, Jagim AR, Jager R, Purpura M, Kerksick CM. Effects of daily 24-gram doses of rice or whey protein on resistance training adaptations in trained males. J Int Soc Sports Nutr. 2020 Dec 1;17(1):60. doi: 10.1186/s12970-020-00394-1. PMID 33261645